CLINICAL TRIAL: NCT05591508
Title: Ketogenic Diet for Status Epilepticus in Infants, Children and Adolescents Aged 6 Months to 18 Years Immediately After Cessation of Convulsive Status Epilepticus; a Randomized Open Labelled Trial
Brief Title: Ketogenic Diet for Status Epilepticus in Children Post Cessation of Convulsive Status Epilepticus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor Sheffali Gulati , Department of Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-140/06.03.2020
Record Dates: First submitted 2022-10-16; First posted 2022-10-24 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Status Epilepticus; Ketogenic Dieting
MeSH Terms: conditions — Status Epilepticus | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Open labeled randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, Intervention Arm (Experimental): Ketogenic Diet +Standard care of Status epilepticus according to current guideline of management
  Interventions: Dietary Supplement: Ketogenic Diet
- B, No Intervention Arm (No Intervention): Standard care of Status Epilepticus according to current guidelines of management

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — Ketogenic diet will be in the form of artificial powder which can be diluted and given through NG tube. It will be started at a ratio of 1:1 followed by daily increment (2:1,3:1 and 4:1) till a urine ketone of 2+ is seen
  Arms: A, Intervention Arm

SUMMARY:
Ketogenic diet being started early in those with status epilepticus and frequent or abundant discharges in EEG in comparison to just standard therapy is being evaluated here for efficacy and adverse effects.

DETAILED DESCRIPTION:
Study Title : Ketogenic diet for status epilepticus in infants, children and adolescents aged 6 months to 18 years immediately after cessation of convulsive status epilepticus; a randomized open labelled trial Objective of The study : To evaluate the efficacy of add on ketogenic diet therapy compared to standard treatment and care of infants, children and adolescents aged 6 months to 18 years in terms of time taken for reduction in EEG discharges by >50% (with a baseline of abundant or frequent discharges) after stoppage of convulsive status epilepticus Justification of the study: Up to one third of epilepsy are medically intractable, of which only another third is surgically amenable. Ketogenic diet is now an established modality of treatment in these 20 percent of patients with epilepsy. Various studies have shown at least up to 50% reduction in seizure frequency with this modality.

The last decade has seen ketogenic diet being used for management of status epilepticus. Current evidence is only in the form of case series and isolated case reports. Status epilepticus is associated with significant mortality and morbidity. Aggressive management is imperative. However, non-convulsive electrographic status may persist beyond cessation of clinical status in up to 20-30% of cases. Thus in such scenarios, it is controversial whether to continue aggressive management with anesthetics and numerous antiepileptics, as the effect may be detrimental. Thus, the current study has been planned to evaluate efficacy of ketogenic diet in status epilepticus.

Study design: Open labeled randomized controlled trial Study population: Infants, children and adolescents aged 6 months to 18 years with electrographic evidence of seizure activity with abundant or frequent discharges immediately after stoppage of convulsive status epilepticus, attending pediatric inpatient services at AIIMS, New Delhi Assuming time to cessation of reduction of EEG discharges by > 50% to be 10+5 days in the KD arm and 15+5 in the non KD arm, with an alpha of 5% and power of 90%, the sample size comes out to be 22 in each arm. It is being proposed that 25 cases will be recruited in each of the arms.

Inclusion criteria

1. Infants, children and adolescents aged 6 months to 18 years
2. Electrographic evidence of seizure(frequent or abundant discharges in EEG)
3. Clinical status controlled immediately on standard therapy and care based on established consensus guidelines followed globally Exclusion criteria

<!-- -->

1. Circulatory failure
2. GI Intolerance
3. Associated chronic systemic illness
4. Any abnormality on baseline laboratory investigation
5. Neurometabolic disorders (except those in which ketogenic diet is therapy of choice)Up to one third of epilepsy are medically intractable, of which only another third is surgically amenable. Ketogenic diet is now an established modality of treatment in these 20 percent of patients with epilepsy. Various studies have shown at least up to 50% reduction in seizure frequency with this modality.

The last decade has seen ketogenic diet being used for management of status epilepticus. Current evidence is only in the form of case series and isolated case reports. Status epilepticus is associated with significant mortality and morbidity. Aggressive management is imperative. However, non-convulsive electrographic status may persist beyond cessation of clinical status in up to 20-30% of cases. Thus in such scenarios, it is controversial whether to continue aggressive management with anesthetics and numerous antiepileptics, as the effect may be detrimental. Thus, the current study has been planned to evaluate efficacy of ketogenic diet in non-convulsive electrographic status.

Study design: Open labeled randomized controlled trial Study population: Infants, children and adolescents aged 6 months to 18 years with electrographic status epilepticus immediately after stoppage of convulsive status epilepticus, attending Pediatric Intpatient services at All India Institute of Medical Sciences (AIIMS), New Delhi Sample size calculation Assuming time to cessation of electrographic status to be 10+-5 days in the KD arm and 15+-5 in the non KD arm, with an α of 5% and power of 90%, the sample size comes out to be 22 in each arm. It is being proposed that 25 cases will be recruited in each of the arms.

Inclusion criteria

1. Infants, children and adolescents aged 6 months to 18 years
2. Electrographic status
3. Clinical status controlled immediately on standard therapy and care based on established consensus guidelines followed globally Exclusion criteria

1. Circulatory failure 2. GI Intolerance 3. Associated chronic systemic illness 4. Any abnormality on baseline laboratory investigation 5. Neurometabolic disorders (except those in which ketogenic diet is therapy of choice) Baseline Assessment The components of baseline assessment of patients are

1. EEG within 6 hours of cessation of clinical status
2. The components of laboratory evaluation will be

   • Complete blood count with peripheral smear with RBC indices

   • Renal and Liver function tests

   • Serum sodium, potassium

   • Fasting blood sugar

   • Serum total protein and albumin

   • Serum calcium, phosphate, alkaline phosphatase

   • Serum lipid profile

   • Venous blood gas

   • Serum uric acid

   • Urine Calcium/creatinine ratio

   • Arterial lactate

   • Serum ammonia

   • Urine GCMS

   • Blood TMS The last 4 investigations will be done if underlying neurometabolic condition is suspected.

Randomisation technique Computer generated block randomization will be done to allocate two groups A and B. Group A will be Add on ketogenic diet therapy + standard care and group B will be only Standard Care.Allocation concealment will be done using sealed envelopes Intervention

1. Setting: In patient services in the Department of Pediatrics, AIIMS, New Delhi
2. Duration: If no improvement is seen within 2 weeks of initiation of ketogenic diet, the therapy will be discontinued. However, in case of response, it will be continued for atleast 4 weeks and then it will be left to the family whether to continue ketogenic diet further or not.
3. Type of intervention: Standard of care therapy will be delivered in both the arms. Add on ketogenic diet therapy will be given to one arm.

   Standard of Care Therapy The standard of care therapy for status epilepticus will be given to patients according to the established global consensus guidelines.

   Dietary therapy will be given for atleast 4 weeks in responders. After baseline investigations, if no contraindication exists, ketogenic diet will be started at the earliest. Ketogenic diet will be in the form of artificial powder which can be diluted and given through NG tube. It will be started at a ratio of 1:1 followed by daily increment (2:1,3:1 and 4:1) till a urine ketone of 2+ is seen.

   The laboratory parameters will be repeated weekly twice on dietary therapy. In case of any abnormality in these investigations, standard established protocol will be followed for management.[84] The tests may be performed more frequently if the clinical condition of the patient demanded so.

   All the patients will be started on oral calcium, levocarnitine (50mg/kg/day, maximum1 gm)and multivitamin tablets.

   Families which opt to continue dietary therapy beyond 4 weeks, standard established protocol will be followed.

   Statistical analysis Baseline variables will be appropriately recorded as continuous or discrete. Comparison between the 2 groups will be done using appropriate bivariate analysis.

   Timelines

   • Enrolment of patients: 0 to 24months

   • Intervention and follow up: 0 to 25 months

   • Data analysis: 25 to 30 months

   .

1. Data management and statistical analysis Data recording would be done in a Microsoft Excel spreadsheet (Microsoft Office, Microsoft Corp., Seattle, WA, USA).

Descriptive: Mean/Median/Range/Standard Deviation/Frequencies would be used to describe the demographic profile of participants and their comorbidities

Categorical variables would be compared using chi square/ Fischer's test Depending upon the distribution of continuous variables Student t test would be used for parametric variables Mann Whitney U test would be used for nonparametric variables. Differences with p value of 0.05 or lower will be considered significant

Ethical aspects Ethical clearance:- The study will be conducted after obtaining Ethical clearance from the Institute Ethical Committee Essentiality and Justification for the study: This study will not only provide unifying insights into multiple aspects of autism, with attendant beneﬁts for improving diagnosis and therapy but also help in bringing this special kind of children/adults to mainstream society.

Consent:- Patients will be enrolled only after obtaining informed written consent from the parents/guardians.

Privacy and confidentiality :- Confidentiality of the records will be maintained

The parents/guardians will have full authority to enroll or withdraw the child from the study and this will not affect the future care and treatment given to the child in our hospital.

Costs of the tests- It will be borne by ICMR, DST, DBT Welcome trust

6.5. Study design: Open labelled randomized controlled trial

6.6 Dosages of drug: Ketogenic diet will be in the form of artificial powder which can be diluted and given through NG tube. It will be started at a ratio of 1:1 followed by daily increment (2:1,3:1 and 4:1) till a urine ketone of 2+ is seen.

6.7 Duration of treatment: Dietary therapy will be given for at least 4 weeks in responders. After baseline investigations

6.8 Investigation: The components of baseline investigations of patients are

1. EEG within 6 hours of cessation of clinical status
2. The components of laboratory evaluation will be • Complete blood count with peripheral smear with RBC indices • Renal and Liver function tests • Serum sodium, potassium • Fasting blood sugar • Serum total protein and albumin • Serum calcium, phosphate, alkaline phosphatase • Serum lipid profile

   • Venous blood gas

   • Serum uric acid

   • Urine Calcium/creatinine ratio

   • Arterial lactate
   * Serum ammonia
   * Urine GCMS
   * Blood TMS The last 4 investigations will be done if underlying neurometabolic condition is suspected.

ELIGIBILITY:
Inclusion Criteria:

1. Infants, children and adolescents aged 6 months to 18 years
2. Electrographic status
3. Clinical status controlled immediately on standard therapy and care based on established consensus guidelines followed globally

Exclusion Criteria:

1. Circulatory failure
2. GI Intolerance
3. Associated chronic systemic illness
4. Any abnormality on baseline laboratory investigation
5. Neurometabolic disorders (except those in which ketogenic diet is therapy of choice)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Ketogenic diet for electrographic status epilepticus in infants, children and adolescents aged 6 months to 18 years immediately after cessation of convulsive status epilepticus; a randomized open labelled trial | 30 Months
  To evaluate the efficacy of add on ketogenic diet therapy compared to standard treatment and care in infants, children and adolescents aged 6 months to 18 years in terms of time taken (in days) for cessation of electrographic status epilepticus immediately after stoppage of convulsive status epilepticus.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Sheffali Gulati, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No